CLINICAL TRIAL: NCT06292741
Title: Evaluation of the Prevalence of Autonomic Nervous System Involvement in Patients With Cognitive Impairment by a Non-invasive Combined Study of Dysautonomia
Brief Title: Autonomic Involvement in Patient With Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4956
Record Dates: First submitted 2023-03-02; First posted 2024-03-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Dementia, Mild; Dementia of Alzheimer Type
MeSH Terms: conditions — Dementia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cognitive decline (Experimental): comparison of autonomic parameters among subjects with different forms of cognitive decline
  Interventions: Device: Sudoscan

INTERVENTIONS:
Device: Sudoscan — recording of sudomotor function and pupillary reactivity
  Other Names: automated pupillometry NPI-200

SUMMARY:
Prospective interventional study with a device for comparing autonomic parameters among patients with different forms of cognitive decline

ELIGIBILITY:
Inclusion Criteria:

* male and females between 50 and 85 years
* cognitive decline (dementia, lewy's body dementia, Parkinson dementia, Alzheimer dementia)
* mild cognitive decline ( lewy's body MCI, Parkinson MCI and Alzheimer MCI)
* Ability to assume the upright position

Exclusion Criteria:

* diabetes mellitus
* eye problems
* severe cognitive decline
* heart disease
* peripheral neuropathy
* language barrier
* oncological disease
* medical pathologies associated with cognitive deficits

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of the prevalence in autonomic dysfunction in patients with MCI and dementia | baseline through study completion, an average of 3 year
  evaluation of the prevalence in autonomic dysfunction in patients with MCI and dementia

SECONDARY OUTCOMES:
correlation between the extent of autonomic involvement and the severity of cognitive decline | baseline through study completion, an average of 3 year
  correlation between the extent of autonomic involvement (pupillary dilatation velocity) and the severity of cognitive decline (MMSE score)
evaluation of the type of cognitive disorder, defined by the scores obtained in the MMSE between subjects with and without autonomic dysfunction. | baseline through study completion, an average of 3 year
  evaluation of the type of cognitive disorder between subjects with and without autonomic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Marra, MD, Principal Investigator — Memory clinic- Policlinico Agostino Gemelli, IRCCS, Università Cattolica del Sacro Cuore I
Locations (1):
- Clinica della memria- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Lazio, Italy